CLINICAL TRIAL: NCT00000263
Title: Effects of Combined Alcohol and Nitrous Oxide Intake
Brief Title: Effects of Combined Alcohol and Nitrous Oxide Intake - 15
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double
Other Study IDs: NIDA-08391-15; R01DA008391 (NIH); R01-08391-15
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Opioid-Related Disorders; Substance-Related Disorders
Keywords: nitrous oxide; ethanol; drug interaction; subjective effects; healthy volunteer
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Nitrous Oxide; Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (3):
- 0 g/Kg ethanol +/- 30% nitrous oxide (Placebo Comparator)
  Interventions: Drug: 30% Nitrous oxide; Other: 0 g/Kg ethanol
- 0.25 g/Kg ethanol +/- 30% nitrous oxide (Active Comparator)
  Interventions: Drug: 30% Nitrous oxide; Other: 0.25 g/Kg ethanol
- 0.5 g/Kg ethanol +/- 30% nitrous oxide (Active Comparator)
  Interventions: Drug: 30% Nitrous oxide; Other: 0.5 g/KG ethanol

INTERVENTIONS:
Drug: 30% Nitrous oxide
Other: 0.25 g/Kg ethanol
  Arms: 0.25 g/Kg ethanol +/- 30% nitrous oxide
Other: 0.5 g/KG ethanol
  Arms: 0.5 g/Kg ethanol +/- 30% nitrous oxide
Other: 0 g/Kg ethanol
  Arms: 0 g/Kg ethanol +/- 30% nitrous oxide

SUMMARY:
The purpose of this study is to determine the effects of combined alcohol and nitrous oxide intake on mood, psychomotor performance, and the pain response in healthy volunteers.

ELIGIBILITY:
Please contact site for information.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 1997-01; Primary Completion 1998-10 (Actual); Study Completion 1998-10 (Actual)

PRIMARY OUTCOMES:
Pain intensity, pain bothersomeness | Post inhalation
Mood | Post inhalation
Psychomotor performance | Post inhalation
Cognitive performance | Post inhalation

CONTACTS AND LOCATIONS:
Overall Officials: James Zacny, Ph.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Anesthesia & Critical Care, Chicago, Illinois, United States